CLINICAL TRIAL: NCT01937260
Title: An Open-label Study to Evaluate the Effect of Brodalumab on the Pharmacokinetics of Midazolam and Assess Single-Dose Brodalumab Pharmacokinetics in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Brodalumab Drug-Drug Interaction (DDI) and Intensive Pharmacodynamic (PK) Study in Psoriasis Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20110184
Record Dates: First submitted 2013-07-15; First posted 2013-09-09 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brodalumab 140mg SC (Experimental): open label, all subjects receive brodulamab
  Interventions: Drug: Brodalumab
- Midazolam (MDZ) 2mg oral, Brodalumab 210mg SC (Experimental): MDZ 2mg oral (Day 1 and Day 9), Brodalumab 210mg SC (Day 2)
  Interventions: Drug: Brodalumab

INTERVENTIONS:
Drug: Brodalumab — Group 1 consists of 20 subjects and will receive 2 oral doses of midazolam and a single SC dose of brodalumab. Group 2 consists of 10 subjects and will receive a single SC dose of brodalumab.
  Other Names: AMG 827

SUMMARY:
This is a phase 1, multi-center, open-label, drug-drug interaction (DDI) and PK study in subjects with moderate to severe plaque psoriasis. It is designed to evaluate the effect of brodalumab on midazolam PK in addition to assessing single dose PK of brodalumab in subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
Approximately 30 subjects will be enrolled into two groups. Group 1 consists of 20 subjects and will receive 2 oral doses of midazolam and a single subcutaneous (SC) dose of brodalumab. Group 2 consists of 10 subjects and will receive a single SC dose of brodalumab.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had stable moderate to severe plaque psoriasis for at least 6 months
* body mass index (BMI) between ≥ 18.0 and ≤ 38.0 kg/m2
* body weight between ≥ 50 and ≤ 130 kg
* no known history of active tuberculosis

Exclusion Criteria:

* Female subjects who are lactating/breastfeeding
* History or evidence of clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- United States (5):
  - Research Site, Anaheim, California
  - Research Site, Irvine, California
  - Research Site, Ocala, Florida
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
- Australia (3):
  - Research Site, Herston, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Prahran, Victoria
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Grafton, Auckland

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Midazolam (MDZ) 2mg Oral (Day 1 and Day 9) Brodalumab 210 mg SC (Day 2)
- Cohort 2: Brodalumab 140 mg SC (Day 1)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 21 | 10
Completed | 20 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Midazolam (MDZ) 2mg oral (Day 1 and Day 9) Brodalumab 210mg SC (Day 2)
- Cohort 2: Brodalumab 140mg SC (Day1)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 10 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (10.9) | 46.8 (15.6) | 43 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 16 | 8 | 24
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Observed Concentration of Midazolam After a Single Dose of Brodalumab
Description: Midazolam pharmacokinetic parameter estimates after single oral dose of Midazolam 2 mg on Day 1 and Day 9 and a single administration of Brodalumab 210 mg on Day 2 with PK sampling collected on Day 30
Time Frame: Day 1 to day 9
Population: Analysis population is now 20 subjects after 1 subject was discontinued by sponsor decision
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
nanograms per milliliter | 11.5 (4.59)

2. Primary Outcome: The Area Under Drug Concentration Time Curve From Zero to Infinity (AUCinf)
Description: as for outcome 1
Time Frame: Day 1 to Day 9
Population: 20 subjects analyzed after the discontinuation of 1 subject by sponsor decision
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Cohort 1: Midazolam (MDZ) 2mg oral (Day 1 and Day 9)Brodalumab 210mg SC (Day 2)
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
hr*ng/mL | 41.5 (22.1)

3. Primary Outcome: The Area Under the Drug-concentration Curve of Midazolam After a Single Dose of Brodalumab From Zero Tot he Last Time of Quantifiable Concentration
Description: Midazolam pharmacokinetic parameter estimates after single oral dose of Midazolam 2 mg on Day 1 and Day 9 and a single administration of Brodalumab 210 mg on Day 2
Time Frame: Day 1 to Day 9
Population: 20 subjects are now analyzed after the discontinuation of 1 subject by sponsor decision
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
hr*ng/mL | 39 (19.2)

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 13/20 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=20) | Cohort 2 (N=10)
Crohn's Disease (Gastrointestinal disorders) | 0 | 1
Injection Site reaction (General disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Muscle Strain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 2 | 0
presyncope (Nervous system disorders) | 1 | 0
headache (Nervous system disorders) | 1 | 0
Catheter Site Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Infected Bites (General disorders) | 1 | 0
Upper Respiratory Tract Infection (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Palpatations (Cardiac disorders) | 1 | 0
Ear Congestion (Ear and labyrinth disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other